CLINICAL TRIAL: NCT06209723
Title: Effect of a Vegetarian Diet on Innate Immunity in Patients With Myocardial Infarction and in Healthy Volunteers (FRESH-MI Study)
Brief Title: Vegetarian Diet and Innate Immunity in Patients With Myocardial Infarction and in Healthy Volunteers (FRESH-MI Study)
Acronym: FRESH-MI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Robin Nijveldt, Prof. dr., Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL84172.091.23
Record Dates: First submitted 2023-07-10; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Diet, Vegetarian

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vegetarian diet (Experimental): Vegetarian diet during five weeks
  Interventions: Other: Vegetarian diet
- No change diet (No Intervention): The 'habitual' diet during five weeks. There are no specific restrictions to their diet.

INTERVENTIONS:
Other: Vegetarian diet — Participants will follow a vegetarian diet during a period of five weeks
  Arms: Vegetarian diet

SUMMARY:
The goal of this clinical trial is to assess the effect of a vegetarian diet on innate immunity of patients with a recent acute myocardial infarction and healthy participants. Also, we will assess the willingness to adapt a more vegetarian eating habit. Study subjects will follow a vegetarian diet for five weeks, whereafter a stabilisation period of six weeks will follow. Then, participants will follow to the other dietary intervention for five weeks. Blood will be drawn at given time points to analyse inflammatory parameters.

DETAILED DESCRIPTION:
We will perform a proof-of-concept study according to a prospective randomized open label blinded endpoint (PROBE) design. Patients with an acute myocardial infarction (AMI) and their healthy life partners / spouses will be randomly assigned to an immediate vegetarian diet or their habitual diet. Patients with AMI will be stratified for non-ST-elevation myocardial infarction (NSTEMI) or ST-elevation myocardial infarction (STEMI). The dietary intervention will start one week after the index event and will comprise a period of five weeks. After a stabilisation phase (six weeks), to assure normalisation of the inflammatory response secondary to the acute myocardial infarction, patients and their spouses will follow the other dietary intervention arm. Then, half of them will start directly with the other dietary intervention and half of them will start after a period of five weeks. Blood samples will be taken at the time points. Also, all participants will be asked to complete a questionnaire at baseline, after twelve weeks and at nine months follow-up. Infarct size as assessed by Cardiovascular Magnetic Resonance (CMR) imaging will be used to adjust cytokine levels.

ELIGIBILITY:
Inclusion Criteria for patients:

* Acute myocardial infarction (STEMI/NSTEMI) with a clear culprit lesion on angiography and successful primary percutaneous coronary intervention (PCI) <1 week before randomisation
* Body mass index between 18.5 and 35 kg/m2
* Written informed consent

Inclusion Criteria for healthy volunteers (life partners / souses)

* Body mass index between 18.5 and 35 kg/m2
* Written informed consent

Exclusion Criteria for patients and healthy volunteers:

* Already on a vegetarian or vegan diet
* Previous myocardial infarction
* Diabetes Mellitus
* Medical history of any disease associated with immune deficiency (either congenital or acquired, including chemotherapy, chronic steroid use, organ transplant)
* Use of immunomodulatory drugs
* Vaccination less than one month before start of intervention
* Clinically significant infections within 1 months prior to start of intervention (defined as fever >38.5 degrees Celsius)
* Active malignant haematological disease
* Known eating disorder (e.g., Anorexia nervosa, Bulimia nervosa)

Exclusion Criteria for healthy volunteers

- Use of lipid lowering therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-08 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
The difference in cytokine production capacity (including TNF-α, IL-6, IL-10, IL-1β) of isolated peripheral blood mononuclear cells (PBMCs) after ex-vivo stimulation before and after the vegetarian diet compared to the habitual diet in patients with AMI | five weeks

SECONDARY OUTCOMES:
The cytokine production capacity (including TNF-α, IL-6, IL-10, IL-1β) of isolated peripheral blood mononuclear cells after ex-vivo stimulation before and after following a vegetarian diet in participants without cardiovascular history. | five weeks
The frequency of the consumption of vegetables per week at nine months follow-up will be compared between patients with a recent acute myocardial infarction, who directly start with a vegetarian diet compared to a deferred start. | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Robin Nijveldt, MD, PhD, Principal Investigator — Radboud University Medical Center; Saloua El Messaoudi, MD, PhD, Study Chair — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
No individual participant data will be shared. Results will be published by the investigators in academic journals. Sharing of generated study data will be carried out in several different ways. We plan to make our results available to researchers and potential collaborators.
Supporting Information: Study Protocol, SAP